CLINICAL TRIAL: NCT07295340
Title: Application of Folic Acid-Targeted Near-Infrared-II (NIR-II) Carbon Dots in Ex Vivo Histopathological Analysis of Hepatocellular Carcinoma
Brief Title: Diagnostic Accuracy of Folate-Targeted NIR-II Carbon Dots for Ex Vivo HCC Detection
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiwei Huang, Clinical Professor, West China Hospital
Other Study IDs: JHuang20234
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Liver Cancer
Keywords: liver cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — resected liver specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group: Patients undergoing standard curative hepatectomy for HCC. Their resected tumor specimens will be used for ex vivo fluorescence imaging analysis.
  Interventions: Diagnostic Test: Ex Vivo FA-CDots Staining

INTERVENTIONS:
Diagnostic Test: Ex Vivo FA-CDots Staining — The resected liver specimens are incubated with Folate-targeted Near-Infrared II Carbon Dots (FA-CDots) and imaged using a NIR-II fluorescence imaging system to identify tumor margins and micro-lesions. The results are compared with standard histopathology.

SUMMARY:
This prospective, single-center observational study evaluates the diagnostic accuracy of a novel Folate-targeted Near-Infrared II Carbon Dot (FA-CDots) probe for the ex vivo assessment of Hepatocellular Carcinoma (HCC). Following standard radical hepatectomy, resected liver specimens will be incubated with the FA-CDots probe and imaged using a NIR-II fluorescence system. The study aims to determine the feasibility and accuracy of this technology in identifying tumor margins and micro-lesions by comparing the fluorescence imaging results with standard histopathological examination.

ELIGIBILITY:
Inclusion Criteria:

1. Primary diagnosis of Hepatocellular Carcinoma (HCC) confirmed clinically or by preoperative biopsy.
2. Scheduled for radical hepatectomy.
3. Preoperative imaging (CT/MRI) suggests indistinct tumor boundaries, infiltrative growth, or proximity to major vessels (expected margin < 1cm).
4. Liver function classified as Child-Pugh Grade A.
5. ASA Physical Status classification I-III.
6. Participant or legal guardian willing to sign informed consent for the use of ex vivo tissues.

Exclusion Criteria:

1. Concomitant other malignant tumors.
2. Severe dysfunction of heart, lung, kidney, or brain unable to tolerate surgery.
3. Recurrent HCC.
4. Preoperative evidence of extrahepatic metastasis or major vascular invasion.
5. Received preoperative anti-tumor therapy.
6. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 diagnosed with hepatocellular carcinoma (HCC) who are scheduled for radical hepatectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance of FA-CDots (Sensitivity, Specificity, and AUC) | Immediate ex vivo analysis post-surgery
  Evaluate the accuracy of FA-CDots in distinguishing HCC tissue from normal liver tissue.
  Metric: Area Under the Receiver Operating Characteristic Curve (AUC), Sensitivity, and Specificity.
  Calculation: Based on the Signal-to-Background Ratio (SBR) of the fluorescence images. A "Positive" result is defined as an SBR > 2.0 (threshold to be optimized).
  Gold Standard: The diagnosis is verified by standard histopathological examination (H&E staining) of the corresponding tissue sites.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No